CLINICAL TRIAL: NCT06767423
Title: Comparative Effectiveness of Targeted Outreach With an Automated Caller for Increasing Appointment Completion: A Randomized Quality Improvement Initiative
Brief Title: Comparing the Effectiveness of Different Appointment Reminder Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M. Kit Delgado, MD (Other)
Responsible Party: Sponsor-Investigator, M. Kit Delgado, MD, Associate Professor of Emergency Medicine, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB # 855257
Record Dates: First submitted 2024-11-13; First posted 2025-01-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Appointment Reminders
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Message (Usual Care) (No Intervention): Standard text message appointment reminders to English and Spanish-speaking patients. Text reminders will go out 3-weeks, 3 days, and 24 hours before the appointment.
- Text Message + Automated Caller (Intervention) (Active Comparator): Standard text message appointment reminders to English and Spanish-speaking patients. Text reminders will go out 3-weeks, 3 days, and 24 hours before the appointment. If patient has not confirmed their appointment after the 3-week and 3-day reminders, they'll receive an automated caller.
  Interventions: Behavioral: Text Message + Automated Caller (Intervention)

INTERVENTIONS:
Behavioral: Text Message + Automated Caller (Intervention) — Standard text message appointment reminders to English and Spanish-speaking patients. Text reminders will go out 3-weeks, 3 days, and 24 hours before the appointment. If patient has not confirmed their appointment after the 3-week and 3-day reminders they will receive an automated caller.
  Arms: Text Message + Automated Caller (Intervention)

SUMMARY:
Penn Medicine is continually trying to optimize operations and decrease number of patients who do not show up for their appointments. This has included new changes to text message reminders, implemented as usual care. At a baseline, less than 75% of scheduled outpatient appointments are actually completed. This results in longer wait times and decreased access for patients and operational inefficiencies. The goal of the project is to test whether supplementing standard text message appointment reminders with targeted outreach using an automated phone call to patients with increased risk of not showing up for their appointment (>15% per Epic's Risk of Patient No-Show Model) reduces no show rate (the study's primary outcome) and increases patient appointment completion rate (% of appointments that were completed during scheduled appointment time, a secondary outcome). Participants will be randomized in a 1:1 ratio to receive either the standard text message or standard text message plus the automated caller. Eligible patients have already consented to receiving text message reminders from Penn Medicine and must have an in-person appointment scheduled during the study period. The Access Optimization Group at Penn will be monitoring the randomization and outcomes reporting of whether a patient confirmed, cancelled, or no showed at the scheduled appointment. All eligible outpatient appointments over a two week period will be included in this operational evaluation. The Access Optimization Group will then make a decision on which approach to implement as usual care based on the results of this operational evaluation.

ELIGIBILITY:
Inclusion Criteria:

* in-person appointments
* English or Spanish speakers
* 18 years old or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32925 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
No Show Rate | Through study completion, on average of 3 weeks
  Proportion of initially scheduled appointments in which the patient did not show.

SECONDARY OUTCOMES:
Appointment Completion Rate | Through study completion, on average of 3 weeks
  Proportion of initial scheduled appointments completed.
Appointment Cancelation Rate | Through study completion, on average of 3 weeks
  Proportion of initially scheduled appointments cancelled.
Appointment Refill Rate | Through study completion, on average of 3 weeks
  Proportion of cancelled appointments that were refilled.
Refilled Appointment Completion Ration | Through study completion, on average of 3 weeks
  Proportion of refilled appointments that were completed.
Net Appointment Completion Rate | Through study completion, on average of 3 weeks
  Proportion of appointment slots resulting in a completed appointment. Includes completed refilled appointments.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Tarabichi Y, Higginbotham J, Riley N, Kaelber DC, Watts B. Reducing Disparities in No Show Rates Using Predictive Model-Driven Live Appointment Reminders for At-Risk Patients: a Randomized Controlled Quality Improvement Initiative. J Gen Intern Med. 2023 Oct;38(13):2921-2927. doi: 10.1007/s11606-023-08209-0. Epub 2023 May 1. PMID 37126125
- See also: Helping Patients Make It to Their Appointments Using Predictive Analytics and Personalized Phone Calls — https://www.epicshare.org/share-and-learn/metrohealth-no-show-predictive-model